CLINICAL TRIAL: NCT04149301
Title: Exploration of the Role of Subtalar Joint Morphology in the Development of Foot Deformity in Cerebral Palsy
Brief Title: Subtalar Joint Morphology and Foot Deformity in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Keele University (Other); Imperial College London (Other); University of Oxford (Other); University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: RL1795
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: musculoskeletal modelling; gait analysis
MeSH Terms: conditions — Cerebral Palsy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Typically developing children: Children who do not have a problem with their walking ie children who do not have cerebral palsy
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: MRI scan
- Children with cerebral palsy without foot deformity
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: MRI scan
- Children with cerebral palsy with mild foot deformity
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: MRI scan
- Children with cerebral palsy with severe foot deformity
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: 3D gait analysis — Children will have their walking measured in the gait laboratory to record their kinematics and kinetics along with electromyography (EMG) from key muscle groups.
Diagnostic Test: MRI scan — The children will have two MRI scans taken - one with the foot loaded and one with no load applied.

SUMMARY:
Cerebral palsy (CP) is a major cause of disability. Many children with CP develop foot deformities as they grow and these can become painful, adversely affecting their quality of life. The research team has previously studied foot morphology and biomechanics, including analysis of the subtalar joint and has successfully located the joint axis from MRI scans.

In this project 25 children will be recruited (15 children with CP and 10 unimpaired control subjects). Each child will attend for a single visit, when they will undergo an MRI scan (with the foot loaded and unloaded) to measure the morphology of the ankle and foot, in particular the subtalar axis alignment. This has not been done before in CP.

Each child will have an instrumented gait analysis and musculoskeletal modelling techniques will be used to study the biomechanical action of the external ground reaction force and internal muscle forces. The potential of these forces to rotate the subtalar joint and deform the foot will be assessed, resulting in new insights into potential mechanisms of foot deformity.

The children will then be categorised to identify those most at risk, leading to personalised screening measures and treatment strategies in the future.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a common cause of childhood disability with an incidence of 2.11 per 1000 live births. Children with CP often develop problems with their feet during growth, with a reported prevalence of foot deformity of 86% in a group of 66 diplegic children. Deformities may occur in the ankle joint, subtalar joint (the joint below the ankle) and/or the foot itself. The European SPARCLE study reported that 54% of children with CP experienced pain in the previous week, which was associated with a poorer quality of life. This rose to 75% in a subsequent study of adolescents. The most common place for children to experience pain is in the feet, especially for the more mobile children.

Clinical experience is that deformed feet are challenging to manage with splints. Biomechanical changes in the ankle and foot affect the whole leg and a sudden deterioration in gait often follows, for example the development of a crouch gait pattern.

Several mechanisms are proposed for the development of foot deformity, including calf muscle tightness, muscle imbalance, bony subluxation and collapse of the longitudinal arch. It is difficult to separate cause and effect as phenomena occur concurrently.

Previously the research team have examined the morphology of the foot in detail using imaging techniques and gait analysis. To date no one has conducted similar studies looking at the subtalar joint in cerebral palsy and the orientation of the axis in this condition is currently unknown.

Participants in this research (typically developing children and children with cerebral palsy) will only need to attend on a single occasion. They will spend around half a day in the hospital, with measurements being taken in two departments:-

MRI scans: The children will have MRI scans taken of one leg. This will be done twice, firstly with the limb unloaded and then with a load applied to the foot. The child will have MRI opaque markers attached to bony landmarks on the skin before the scans are taken.

Gait analysis: The children will attend the gait laboratory. Here they will be asked to wear shorts and a T shirt or crop top. A simple orthopaedic examination will be carried out to measure their legs and joints. They will then have retroreflective markers and electromyography (EMG) sensors attached to their legs and they will be asked to walk up and down the laboratory whilst their walking pattern is recorded. The record will include video images, 3D tracking of the marker positions and muscle signals from the EMG.

At the end of the data collection they will be free to leave and their participation in the study will end.

MRI scans will be segmented using Mimics (Materialise, Belgium) software to obtain bone geometries. As demonstrated in previous studies unloaded MRI scans allow high quality reconstruction of foot bone geometries, suitable for generating multi-segmental models of the foot and tibia in adult and paediatric populations. Subject-specific ankle and foot musculoskeletal models will be produced from the reconstructed patient's bone geometries, including personalized muscle attachments, derived from the MRI scans and subject-specific tibiotalar and subtalar joint axes, identified by fitting appropriate analytical shapes (spheres and cylinders) to the articular surfaces.

The individual dynamic models will be validated by comparing their configuration in the stance phase of walking against the loaded MRI scans. External joint moments due to the action of ground reaction force will be computed using an inverse dynamics analysis implemented in OpenSim, while the contribution of the calf muscles to the internal joint moments will be estimated by computing the muscles' moment arms with respect to foot joint axes.

This study will produce the first pilot data of static and dynamic subtalar morphology in children with cerebral palsy. The research team hope to identify potential mechanisms of deformity which can be used to categorise feet and inform treatment, prior to designing a future interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk independently (for CP children GMFCS level 1 or 2)
* Able to understand and comply with experimental protocols

Exclusion Criteria:

* Any contraindications to MRI scanning eg pronounced startle reflexes or metal implants.
* Any orthopaedic surgery in the last 6 months, or any previous bony surgery to the ankle of foot.

Ages: 7 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children with cerebral palsy and typically developing children aged 7-16 years.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
External loading on the subtalar joint (Measured as a moment in units of Nm) | At baseline
  This results from combining the gait analysis data (angles and forces) with the morphology from the MRI scans.
Internal loading on the subtalar joint (Measured as a moment in units of Nm) | At baseline
  This results from combining the gait analysis data (angles and forces) with the morphology from the MRI scans, through a process of optimisation to distribute internal muscle forces.

CONTACTS AND LOCATIONS:
Locations (1):
- ORLAU, RJAH Orthopaedic Hospital, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data will only be shared within the research team during the research study, though anonymised data may be released with publication.

REFERENCES:
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] O'Connell PA, D'Souza L, Dudeney S, Stephens M. Foot deformities in children with cerebral palsy. J Pediatr Orthop. 1998 Nov-Dec;18(6):743-7. PMID 9821129
- [Background] Parkinson KN, Dickinson HO, Arnaud C, Lyons A, Colver A; SPARCLE group. Pain in young people aged 13 to 17 years with cerebral palsy: cross-sectional, multicentre European study. Arch Dis Child. 2013 Jun;98(6):434-40. doi: 10.1136/archdischild-2012-303482. Epub 2013 Apr 20. PMID 23606716
- [Background] Montefiori E, Modenese L, Di Marco R, Magni-Manzoni S, Malattia C, Petrarca M, Ronchetti A, de Horatio LT, van Dijkhuizen P, Wang A, Wesarg S, Viceconti M, Mazza C; MD-PAEDIGREE Consortium. An image-based kinematic model of the tibiotalar and subtalar joints and its application to gait analysis in children with Juvenile Idiopathic Arthritis. J Biomech. 2019 Mar 6;85:27-36. doi: 10.1016/j.jbiomech.2018.12.041. Epub 2019 Jan 9. PMID 30704761
- [Background] Modenese L, Montefiori E, Wang A, Wesarg S, Viceconti M, Mazza C. Investigation of the dependence of joint contact forces on musculotendon parameters using a codified workflow for image-based modelling. J Biomech. 2018 May 17;73:108-118. doi: 10.1016/j.jbiomech.2018.03.039. Epub 2018 Mar 30. PMID 29673935
- [Background] Parr WC, Chatterjee HJ, Soligo C. Calculating the axes of rotation for the subtalar and talocrural joints using 3D bone reconstructions. J Biomech. 2012 Apr 5;45(6):1103-7. doi: 10.1016/j.jbiomech.2012.01.011. Epub 2012 Jan 28. PMID 22284429
- [Background] Delp SL, Anderson FC, Arnold AS, Loan P, Habib A, John CT, Guendelman E, Thelen DG. OpenSim: open-source software to create and analyze dynamic simulations of movement. IEEE Trans Biomed Eng. 2007 Nov;54(11):1940-50. doi: 10.1109/TBME.2007.901024. PMID 18018689